CLINICAL TRIAL: NCT06112041
Title: The Prospective Clinical Study of Precision PRaG Therapy in Elderly Patients With Advanced Solid Malignant Tumors(PRaG9.0)
Brief Title: The Prospective Clinical Study of Precision PRaG Therapy in Elderly Patients With Advanced Solid Malignant Tumors (PRaG9.0)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JD-LK2023082-I01
Record Dates: First submitted 2023-10-23; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Carcinoma; Solid Tumor
MeSH Terms: conditions — Carcinoma | interventions — Radiotherapy; Thymopentin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADC Combined With Radiotherapy, PD-L1 Sequential GM-CSF and Thymopentin (Experimental): ADC Combined With Radiotherapy, PD-L1 Sequential GM-CSF and Thymopentin
  Interventions: Drug: ADC Combined With Radiotherapy, PD-L1 Sequential GM-CSF and Thymopentin

INTERVENTIONS:
Drug: ADC Combined With Radiotherapy, PD-L1 Sequential GM-CSF and Thymopentin — RC48-ADC combined with hypofractionated radiotherapy, PD-L1 inhibitor sequential GM- CSF and Thymopentin

SUMMARY:
This is an open-label, single-arm, Phase II investigator-initiated trial of hypofractionated radiotherapy combined with PD-L1 inhibitor sequential GM-CSF and thymopentin for treatment of elderly patients with advanced solid tumors, when the HER-2 positive patients are treated with extra antibody-drug conjugate.

ELIGIBILITY:
Inclusion Criteria:

* Aged 75 years and above
* Standard treatment is ineffective (disease progresses after treatment) or locally advanced or metastatic malignant solid tumor patients who cannot tolerate standard therapy, cannot receive or do not have standard therapy
* ECOG(Eastern Cooperative Oncology Group) performance is 0-3
* Life expectancy greater than 3 months
* serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤3.0*ULN, or AST and ALT≤5*ULN with hepatic metastasis; Total serum creatinine ≤1.5*ULN
* Signed informed consent form

Exclusion Criteria:

* Current pregnancy or lactation
* History of other malignant tumors within 5 years prior to dose administration, expect for#malignancies that can be cured after treatment (including but not limited to adequately treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer)
* Uncontrolled epilepsy, central nervous system diseases or mental illness
* arrhythmia, congestive heart failure, or greater than or equal to Class 2 congestive heart failure as defined by the New York Heart Association Functional Classification, or history of myocardial infarction unstable angina, or acute coronary syndrome within 6 months prior to enrollment in the study
* Received allogeneic hematopoietic stem cell transplantation or solid organ transplantation
* Other serious, uncontrolled concomitant diseases that may affect protocol compliance or interpretation of outcomes, including active opportunistic infections or advanced (severe) infections, uncontrolled diabetes
* Allergic to any of the ingredients used in the study
* A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency disease, or a history of organ transplantation, or other immune-related disease requiring long-term oral hormone therapy
* Acute and chronic tuberculosis infection
* Other disorders with clinical significance according to the researcher's judgment

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-10-25 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate #ORR# | 36 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | 36 months
  PFS was defined as the time from the first administration of study treatment to the first occurrence of disease progression as determined by investigator using RECIST v1.1 or death from any cause, whichever comes first.
Disease control rate (DCR) | 36 months
  DCR was defined as the percentage of participants with a complete response (CR), partial response (PR), or stable disease (SD).
Overall survival (OS) | 36 months
  OS was defined as the time from the first administration of study treatment to death from any cause.
Adverse event | 36 months
  rate of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Soochow University, Suzhou, China

REFERENCES:
- [Derived] Zhao X, Yang M, Zhang J, Kong Y, Xu M, Chen R, Yin Q, Wang S, Chen G, Xing P, Zhang L. Efficacy and Safety of PRaG Therapy in Elderly Patients with Advanced Malignant Tumors: A Prospective, Multicenter Clinical Study Protocol (PRaG 9.0 Study). Technol Cancer Res Treat. 2025 Jan-Dec;24:15330338251400412. doi: 10.1177/15330338251400412. Epub 2025 Nov 27. PMID 41308040